CLINICAL TRIAL: NCT06110013
Title: Value of Non Invasive Hemodynamic Monitoring in Patients Admitted to Respiratory Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Sayed Ahmed, Resident doctor, Assiut University
Other Study IDs: Hemodynamic monitoring
Record Dates: First submitted 2023-09-19; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Non-invasive Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- A: Patients on invasive mechanical ventilation
  Interventions: Device: Electrical cardiometry
- B: Patients on Non invasive mechanical ventilation
  Interventions: Device: Electrical cardiometry
- C: Patients Not on mechanical ventilation
  Interventions: Device: Electrical cardiometry

INTERVENTIONS:
Device: Electrical cardiometry — All included patients will be connected to Electrical cardiometry device. The electrodes will be placed over the bare skin of patients at the following sites:
  A. on the left neck below the ear B. directly superior to the midpoint of the left clavicle C. along the left mid-axillary line at the level of the xiphoid process D. two inches below the third electrode. High frequency signals pass through 2 acting electrodes, the other 2 measuring electrodes detect changes in bioimpedance resistance to allow continuous hemodynamic monitoring, then data will be analysed to give comprehensive picture of the hemodynamic circulatory system, allowing differential diagnosis for a patient management
  Other Names: ICON

SUMMARY:
This study aims to evaluate clinical application of electrical cardiometry EC in patients admitted to respiratory ICU. It will evaluate the reliability of EC in assessment of hemodynamic changes in these patients. It will estimate the effect of mechanical ventilation either invasive or non invasive hemodynamic parameters in patients admitted to ICU with respirator disorders

DETAILED DESCRIPTION:
Mechanical ventilation MV is a life saving intervention in intensive care units. Access to lower airways is achieved either through tracheostomy or endotracheal intubation. More recently non invasive ventilation NIV techniques were introduced that do not require an endotracheal airway but using patient ventilator interfaces in the form of facial masks have been designed.

The haemodynamic consequences of MV are multiple and complex and may affect all the determinants of cardiac performance such as heart rate.preload.contractility .and afterload. These consequences affect both right and left ventricle and are also related to the biventricular interdependence .

Mechanically ventilated patients are considered Critically ill.and they are often hemodynamically unstable or at risk of becoming unstable owing to hypovolemia. cardiac dysfunction. or alterations of vasomotor function. leading to organ dysfunction.deterioration into multiorgan failure .and eventually death .Socardiopulmonary monitoring is crucial to ensure successful evaluation and management of these patients . With hemodynamic monitoring. The investigators aim to guide our medical management to prevent or treat organ failure and improve the outcomes of our patients. Therapeutic measures may include fluid resuscitation.vasopressors or inotropic agents .

Hemodynamic monitoring can be done by different techniques which ranges from invasive to less invasive and completely noninvasive methods to assess Cardiac output BP oxygen saturation. Some hemodynamic parameters are easy to be measured like blood pressure and heart rate but do not give a complete picture of a patient's hemodynamics .

Measuring CO and its components preload afterload and contractility will tell us if there is ongoing need for fluid resuscitation vasopressors or inotropic agents . It can be used as a diagnostic tool to determine the type of shock hypovolemic cardiogenic obstructive or distributive according to the hemodynamic profile .

Traditional invasive methods incorporate thermodilution which requires that a transvenous catheter pushed forward to the pulmonary artery PAC Swan Ganz catheter. Other invasive methods require an arterial line to measure the blood pressure signal waveform . Due to the invasiveness the associated risk invasive methods are usually employed at an advanced stage of illness .

Non invasive hemodynamic methods have less complications. Recent techniques advances led to continuous non invasive monitoring that allow for data obtaining at bedside of critically ill patients in ICU these advances help to monitor changes and allow for management before complications .

A portable Electro Cardiometer ICON Osypka Medical GmbH Berlin Germany is a Hand held Portable battery operated non invasive cardiometer for continuous measurement of different hemodynamic parameters stroke volume SV cardiac output CO contractility fluid status and oxygen status in neonate children or adults Applied to the patients through 4 ECG electrodes. It is based on the measurement of changes in thoracic impedance to an electrical current that is produced by fluctuations in thoracic blood volume with each cardiac cycle .

Newer generation Thoracic Electrical Bioimpedence methods have overcome some of the limitations that was present in old models by having faster signal processing better signal filters improved ECG triggering and respiratory filtering .

Up till now there is limited research about ICON device and it's reliability in monitoring hemodynamics specially in respiratory ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to respiratory intensive care unit (ICU) among both sexes Age >18 years Old.

Exclusion Criteria:

1. Patients less than 18 years old .
2. Pregnant women.
3. Patients with injuries, burns, or wounds which precluded the proper application of the device electrodes will be also excluded from the study.
4. those with uncontrollable fits.
5. Patients who need electrical direct current (DC) shock.
6. Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to respiratory intensive care unit (ICU)
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of non invasive hemodynamic monitoring | Baseline
  Effectiveness of clinical application of non invasive hemodynamic monitoring using electrical cardiometer in patients admitted to respiratory intensive care unit

REFERENCES:
- [Result] Masip J. Non-invasive ventilation. Heart Fail Rev. 2007 Jun;12(2):119-24. doi: 10.1007/s10741-007-9012-7. PMID 17492379
- [Result] Russell A, Rivers EP, Giri PC, Jaehne AK, Nguyen HB. A Physiologic Approach to Hemodynamic Monitoring and Optimizing Oxygen Delivery in Shock Resuscitation. J Clin Med. 2020 Jun 30;9(7):2052. doi: 10.3390/jcm9072052. PMID 32629778
- [Result] Nagel JH, Shyu LY, Reddy SP, Hurwitz BE, McCabe PM, Schneiderman N. New signal processing techniques for improved precision of noninvasive impedance cardiography. Ann Biomed Eng. 1989;17(5):517-34. doi: 10.1007/BF02368071. PMID 2610423